CLINICAL TRIAL: NCT03350204
Title: Biomechanical Outcomes Associated With Osteoarthritis Progression in Meniscectomy Patients During Athletic and Functional Tasks (BOOM Study)
Brief Title: Biomechanical Osteoarthritis Outcomes in Meniscectomy Patients
Acronym: BOOM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salford (Other)
Responsible Party: Principal Investigator, Vanessa Walters, Miss, University of Salford
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: HSR1617-56
Record Dates: First submitted 2017-11-17; First posted 2017-11-22 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Meniscus Injury; Meniscectomy; Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Meniscectomy

STUDY DESIGN:
Intervention Model Description: Testing both meniscus patients and uninjured individuals for comparison
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meniscus Injured (Experimental): These participants will come in pre and post operation
  Interventions: Procedure: Meniscectomy
- Healthy (Experimental): These participants will be used as a standardised comparison for the patient group
  Interventions: Other: Helathy control comparison

INTERVENTIONS:
Procedure: Meniscectomy — This will be to see what occurs in both kinetics and kinematics after you have a surgery and how this links on to osteoarthritis
  Arms: Meniscus Injured
Other: Helathy control comparison — This group will be used to get a baseline for normal and natural walking, running and other several tasks which will be used as a comparison for the meniscus injury group.
  Arms: Healthy

SUMMARY:
The key aim of this study is to examine biomechanical measures associated with osteoarthritis (OA) progression in patients who have lateral and medial menisci injuries during various tasks. The likelihood is that individuals who have a meniscal injury often develop knee osteoarthritis. Therefore understanding biomechanical changes from the injury, specifically undertaking both functional and sporting activities, may provide a conservative approach to delaying or minimising the development of OA. Three-dimensional kinetic and kinematic measures will be assessed during seven tasks (walking, running, side cuts, single leg landing, small knee bend squat and isokinetic leg strength), prior to and following treatment. In addition, Strength and balance will be assessed to indicate if there is more work in the rehabilitation program that is needed for functional movement.

DETAILED DESCRIPTION:
Injuries to the meniscus are common in sport, often as a result of a traumatic event (Englund et al., 2016; Stanley et al., 2016; Yeh et al., 2012). Mitchell et al. (2016) reported 5.1 meniscal injuries per 100 000 athletic exposures, with a greater proportion reported during competition (11.9 injuries per 100 000 athletic exposures), compared to practice (2.7 injuries per 100 000 athletic exposures). Rotation around a planted/ inverted foot has been cited as a common mechanism for meniscal injuries, followed by landing and jumping movements. The meniscus aids in stabilising the knee, acting as a shock absorber and transmitting load, with the lateral meniscus taking as much as 70% of the load in the lateral compartment and the medial meniscus carrying approximately 50% of the medial load (Fox et al., 2015; Kurosawa et al., 1980). The lateral meniscus is of particular importance in young active people, especially in athletes and sportsmen. The geometries of the medial and lateral compartments differ significantly (McDermott, 2011).

Damage to the meniscus is suggest to lead to altered knee mechanics leading to the initiation or acceleration of osteoarthritis (OA) development (Badlani et al., 2013; Englund et al., 2016). Prior meniscal tears are commonly reported in OA patients (Bhattacharyya et al., 2003), in addition, reports suggest 4 to 14 times increased risk of developing OA following a meniscal injury (Gelber et al., 2000; Kujala et al., 1995).

Altered knee mechanics have been reported following a meniscal injury, which have been associated with increased likelihood of developing OA, the exact affects differ however depending on which compartment of the meniscus has been operated (Hulet et al., 2014). These changes include reduced contact area within the joint and increased contact pressure, resulting in reduced ability to transmit load (Badlani et al., 2013). Indirect measures of knee loading, such as external knee adductor moments and knee adduction angular impulses (KAAI), have been associated with increased risk of developing OA (Chang et al., 2014). Knee joint loading is also determined by the coordination of muscle activity (Schmitt & Rudolph, 2008). Greater and longer co-contractions of the medial muscles at the knee have demonstrated faster development of OA in individuals diagnosed with medial knee OA (Hodges et al., 2016).

Meniscectomies are widely used to manage the symptoms associated with meniscus injuries (McDermott, 2011). Whilst, non-operative therapies have demonstrated improvements in knee pain three years post intervention (Rimington et al., 2009). However, following these interventions, alter mechanics of the knee have been observed (Badlani et al., 2013; Edd et al., 2015; Willy et al., 2016). For instance, following a medial meniscectomy, increases in contact area and pressure at the knee have been observed and suggested to increase the likelihood of developing OA (Bae et al., 2012). As many athletic individuals with a meniscal lesion undergo partial meniscectomy with the goal of returning to sports participation, knowledge of knee joint loads during such activities are important and under researched and may inform effective rehabilitation measures (Willy et al., 2016). Due to reduced tibiofemoral contact area, a knee that has undergone a partial meniscectomy has a diminished capacity to manage loads (Atmaca et al., 2013). Meniscectomy patients have demonstrated increased external knee adduction moment (EKAM) three months post operation (Hall et al., 2014), this increase could explain the increase risk of OA progression reported in these patients. Medial compartment knee osteoarthritis is often initiated by changes in knee joint motions and increased contact forces, such as those following meniscal injuries. The external knee adduction moment (EKAM) has been identified as a surrogate measure for medial contact force during gait, with an abnormally large peak value being linked to increased pain and rate of disease progression (Walter et al., 2010). The external knee adduction moment Increases in EKAM in meniscectomy patients have been associated with changes in tibia alignment and ground reaction force (GRF) lever arm (Hall et al., 2014; Hunt et al., 2006). Non-invasive interventions such as footwear, could alter biomechanics to lower EKAM and reduce the progression of OA. However, firstly an understanding of the lower limb biomechanics in these individuals is needed Despite the information about contributing factors and underlying mechanisms of meniscus injuries and the progression to OA, there is still a lack in current literature on specific movement patterns, rehabilitation strategies and sport influences. For instance, majority of research examines walking with only Willy et al. (2016) examining running. Typical sports movements such landing and cutting require dynamic control of the knee which is very under-researched (Hall et al., 2015). Muscle strength recovery is also considered to be important for young individuals after an arthroscopic surgery in order to regain capacity to participate in sports or other activities as both pre- and post-operative knee extensor strength have been reported to predict better functional outcome of knee surgery (Pietrosimone et al., 2016). Recent studies that analysed both the peak force and rate to peak force development have shown that there is a significant reduction in muscle strength post meniscectomy treatment (Eitzen et al., 2009). This is considered to be clinically relevant for the return to sport criteria, as most meniscectomy patients have been seen to have a 25% strength difference between legs (Hall et al., 2013), however for patients with knee injuries this difference is often capped at 10% difference between legs to return to their sports (Grindem et al., 2016). Muscle strength is also essential to control movements such as stair descent which is essential for everyday living (Rudolph and Snyder-Mackler., 2004). This is closely linked with balance and the risk of falling. The current literature shows a large variability in assessment methods and results. However, no assessment in isolation can provide a full picture of the problem. A combination of assessment tools seems crucial, since it enables the supply of a full picture meniscus injuries and coping mechanisms. By means of an integrated approach, underlying mechanisms of meniscectomies can be identified, and the adequate treatments such as individualized movements, activity levels and specific shoes can be identified. This should facilitate more informed biomechanical outcomes conveying measures that can be implemented to diminish the risks of OA in meniscectomy patients, in the hopes of improving and aiding their recovery indefinitely.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 40 years
2. Meniscal injury sustained during a sporting task e.g. a sports cutting manoeuvre (Football, Basketball, Netball, Hockey etc.)
3. Compete and or play sport a minimum two times a week
4. Able to perform sport specific tasks including running, single leg landing and small knee bend squat
5. Medial or a lateral meniscal tear and listed for surgery
6. Surgery in the last 12 months for meniscal injury (Meniscectomy or Meniscal Repair)

Exclusion Criteria:

1. History of lower extremity surgeries e.g. ACL reconstruction (other than meniscal injury)
2. Evidence of knee osteoarthritis development either assessed clinically (based on ACR criteria) or radiographically (Kellgren-Lawrence grade >1)
3. Previous history of traumatic (other than the sustained meniscal injury), inflammatory or infectious pathology in the lower extremity
4. Evidence of ligament laxity
5. Degenerative aspects including tear

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-09-20 (Actual); Study Completion 2020-09-20 (Actual)

PRIMARY OUTCOMES:
Biomechanics | Immediate
  All sections of the knee adduction moment curve (different peaks) and also the knee adduction angular impulse (the area under the curve) will be assessed for differences between conditions. Magnitudes and durations of three muscle co-contractions will be calculated from the surface EMG data

SECONDARY OUTCOMES:
Knee injury and osteoarthritis outcome score (KOOS) | Immediate
  The KOOS consists of five subscales; Pain, other symptoms, function in daily living (ADL), function in sport and recreation (Sport/Rec) and knee related quality of life (QOL). A five point Likert scale is employed in the questionnaire, with the last week is taken into consideration when answering the questions. A normalised score is calculated for each subscale with a score of 100 indicting no symptoms, whilst 0 indicates extreme symptoms.
Patient-perceived global change in pain | Immediate
  Patients-perceived global change in pain will be assessed during the tasks. Participants will be asked to complete the five point Likert scale (1 - much worse, 2 - slightly worse, 3 - no change, 4 - slightly better, 5 - much better) following each task (Hinman et al., 2008).
Tampa Scale of Kinesiophobia (TSK) | Immediate
  The TSK is a 17-item questionnaire, which asks individuals to rate the extent to which they agree with statements such as 'pain always means that I injured my body' on a 4-point rating scale, with 1 = strongly disagree and 4 = strongly agree (Nicholas et al., 2008). This is to look at whether any changes in the data are because a participant physically cannot move any different or whether they are subconsciously cautious because they have a fear of pain (Miller, Kori and Todd 1991).

CONTACTS AND LOCATIONS:
Locations (1):
- Manchester Institute of Health and Performance, Manchester, Lancashire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The research data will only be shared in the research team participating in this study.